CLINICAL TRIAL: NCT05997797
Title: Translation, Cross-Cultural Adaptation and Reliability of Urdu Version of The Foot and Ankle Ability Measures (FAAM-U)
Brief Title: Translation and Reliability of FAAM-U
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: IRB- UOL-FAHS/810-XXII/2021
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Foot Injuries; Ankle Injuries
MeSH Terms: conditions — Foot Injuries; Ankle Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group: A total of 175 patients with a range of foot or ankle problems were included for the review. Informed consent was taken from the review members in written form. They all finished the Urdu version of FAAM in the test session. With a time, span of 3 days after the primary recording, a total of the 175 patients whose conditions were relied upon to stay stable were approached to complete the forms again in the retest meeting; no treatment was given during this time-frame. The FAAM is made out of two subscales including ADL and Sports subscales that have a complete score of 84 and 32, individually. Also, toward the finish of the structure, patients were approached to rate the current degree of function with a 4-point Likert scale. Patients evaluated everything as indicated by the trouble they go over with each undertaking on account of their foot or ankle condition. After assortment, information was saved in a safe spot to keep away from any dispositions.
  Interventions: Other: FAAM

INTERVENTIONS:
Other: FAAM — The FAAM is made out of two subscales including ADL and Sports subscales that have a complete score of 84 and 32, individually

SUMMARY:
This study is designed to translate and validate the FAAM questionnaire to the Urdu language, to interpret its psychometric properties, and to determine the reliability of scores obtained from the population of Pakistan. The translated version of the gold standard tool will be used by the local population as well as Urdu-speaking immigrants across the globe to better understand and report the severity of their symptoms. Hence, to improve quality of life across cultures, there is a need of standard outcome measures in Urdu language.

ELIGIBILITY:
Inclusion Criteria:

* Ankle and foot disorders, referred by a general physician or surgeon,
* Conscious
* Ambulatory
* Able to write and read Urdu language

Exclusion Criteria:

* inflammatory disease
* vascular diseases
* neural diseases
* cancer

Ages: 16 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: With a time, span of 3 days after the primary recording, a total of the 175 patients whose conditions were relied upon to stay stable were approached to complete the forms again in the retest meeting; no treatment was given during this time-frame.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
FAAM-U | 72 Hours
  The FAAM is made out of two subscales including ADL and Sports subscales that have a complete score of 84 and 32, individually. Also, toward the finish of the structure, patients were approached to rate the current degree of function with a 4-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Guyatt GH, Sackett DL, Sinclair JC, Hayward R, Cook DJ, Cook RJ. Users' guides to the medical literature. IX. A method for grading health care recommendations. Evidence-Based Medicine Working Group. JAMA. 1995 Dec 13;274(22):1800-4. doi: 10.1001/jama.274.22.1800. No abstract available. PMID 7500513
- [Background] Cervera-Garvi P, Ortega-Avila AB, Morales-Asencio JM, Cervera-Marin JA, Martin RR, Gijon-Nogueron G. Cross-cultural adaptation and validation of Spanish version of The Foot and Ankle Ability Measures (FAAM-Sp). J Foot Ankle Res. 2017 Aug 22;10:39. doi: 10.1186/s13047-017-0221-6. eCollection 2017. PMID 28852426
- [Background] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Martin RL, Irrgang JJ. A survey of self-reported outcome instruments for the foot and ankle. J Orthop Sports Phys Ther. 2007 Feb;37(2):72-84. doi: 10.2519/jospt.2007.2403. PMID 17366962
- [Background] Cuesta-Vargas AI, Gabel CP, Bennett P. Cross cultural adaptation and validation of a Spanish version of the Lower Limb Functional Index. Health Qual Life Outcomes. 2014 May 17;12:75. doi: 10.1186/1477-7525-12-75. PMID 24885123
- [Background] Nelson EC, Eftimovska E, Lind C, Hager A, Wasson JH, Lindblad S. Patient reported outcome measures in practice. BMJ. 2015 Feb 10;350:g7818. doi: 10.1136/bmj.g7818. No abstract available. PMID 25670183
- [Background] Cuesta-Vargas AI, Gabel PC. Cross-cultural adaptation, reliability and validity of the Spanish version of the Upper Limb Functional Index. Health Qual Life Outcomes. 2013 Jul 26;11:126. doi: 10.1186/1477-7525-11-126. PMID 23889883
- [Background] Forget NJ, Higgins J. Comparison of generic patient-reported outcome measures used with upper extremity musculoskeletal disorders: linking process using the International Classification of Functioning, Disability, and Health (ICF). J Rehabil Med. 2014 Apr;46(4):327-34. doi: 10.2340/16501977-1784. PMID 24531349
- [Background] De Noronha M, Refshauge KM, Kilbreath SL, Figueiredo VG. Cross-cultural adaptation of the Brazilian-Portuguese version of the Cumberland Ankle Instability Tool (CAIT). Disabil Rehabil. 2008;30(26):1959-65. doi: 10.1080/09638280701809872. PMID 18720109
- [Background] Martin RL, Hutt DM, Wukich DK. Validity of the Foot and Ankle Ability Measure (FAAM) in Diabetes Mellitus. Foot Ankle Int. 2009 Apr;30(4):297-302. doi: 10.3113/FAI.2009.0297. PMID 19356352
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Bago d'Uva T, Van Doorslaer E, Lindeboom M, O'Donnell O. Does reporting heterogeneity bias the measurement of health disparities? Health Econ. 2008 Mar;17(3):351-75. doi: 10.1002/hec.1269. PMID 17701960
- [Background] Lin CI, Houtenbos S, Lu YH, Mayer F, Wippert PM. The epidemiology of chronic ankle instability with perceived ankle instability- a systematic review. J Foot Ankle Res. 2021 May 28;14(1):41. doi: 10.1186/s13047-021-00480-w. PMID 34049565
- [Background] Lopez-Lopez D, Perez-Rios M, Ruano-Ravina A, Losa-Iglesias ME, Becerro-de-Bengoa-Vallejo R, Romero-Morales C, Calvo-Lobo C, Navarro-Flores E. Impact of quality of life related to foot problems: a case-control study. Sci Rep. 2021 Jul 15;11(1):14515. doi: 10.1038/s41598-021-93902-5. PMID 34267276
- [Background] Saleh, A.M., et al., PSYCHOMETRIC PROPERTIES OF TRANSLATED ARABIC VERSION OF FOOT AND ANKLE ABILITY MEASURE QUESTIONNAIRE. 32: p. 3.
- [Background] Nauck T, Lohrer H. Translation, cross-cultural adaption and validation of the German version of the Foot and Ankle Ability Measure for patients with chronic ankle instability. Br J Sports Med. 2011 Aug;45(10):785-90. doi: 10.1136/bjsm.2009.067637. Epub 2009 Dec 2. PMID 19955163
- [Background] Sartorio F, Vercelli S, Bravini E, Bargeri S, Moroso M, Plebani G, Ferriero G. [Foot and ankle ability measure: cross-cultural translation and validation of the Italian version of the ADL module (FAAM-I/ADL)]. Med Lav. 2014 Jul 15;105(5):357-65. Italian. PMID 25134631
- [Background] Mazaheri M, Salavati M, Negahban H, Sohani SM, Taghizadeh F, Feizi A, Karimi A, Parnianpour M. Reliability and validity of the Persian version of Foot and Ankle Ability Measure (FAAM) to measure functional limitations in patients with foot and ankle disorders. Osteoarthritis Cartilage. 2010 Jun;18(6):755-9. doi: 10.1016/j.joca.2010.03.006. Epub 2010 Mar 23. PMID 20338253
- [Background] Uematsu D, Suzuki H, Sasaki S, Nagano Y, Shinozuka N, Sunagawa N, Fukubayashi T. Evidence of validity for the Japanese version of the foot and ankle ability measure. J Athl Train. 2015 Jan;50(1):65-70. doi: 10.4085/1062-6050-49.3.42. Epub 2014 Oct 13. PMID 25310247
- [Background] Angthong C. Validity and reliability of Thai version of the Foot and Ankle Outcome Score in patients with arthritis of the foot and ankle. Foot Ankle Surg. 2016 Dec;22(4):224-228. doi: 10.1016/j.fas.2015.09.006. Epub 2015 Oct 13. PMID 27810018
- [Background] Gonzalez-Sanchez M, Li GZ, Ruiz Munoz M, Cuesta-Vargas AI. Foot and ankle ability measure to measure functional limitations in patients with foot and ankle disorders: a Chinese cross-cultural adaptation and validation. Disabil Rehabil. 2017 Oct;39(21):2182-2189. doi: 10.1080/09638288.2016.1219772. Epub 2016 Sep 6. PMID 27597231
- [Background] Celik D, Malkoc M, Martin R. Evidence for reliability, validity and responsiveness of Turkish Foot and Ankle Ability Measure (FAAM). Rheumatol Int. 2016 Oct;36(10):1469-76. doi: 10.1007/s00296-016-3485-4. Epub 2016 May 2. PMID 27136921
- [Background] Borloz S, Crevoisier X, Deriaz O, Ballabeni P, Martin RL, Luthi F. Evidence for validity and reliability of a French version of the FAAM. BMC Musculoskelet Disord. 2011 Feb 8;12:40. doi: 10.1186/1471-2474-12-40. PMID 21303520
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Background] Brown, T.A., Confirmatory factor analysis for applied research. 2015: Guilford publications.
- [Background] Andresen EM. Criteria for assessing the tools of disability outcomes research. Arch Phys Med Rehabil. 2000 Dec;81(12 Suppl 2):S15-20. doi: 10.1053/apmr.2000.20619. PMID 11128900
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Maskey, R., et al., Use of exploratory factor analysis in maritime research. 2018. 34(2): p. 91- 111.
- [Background] Arunakul M, Arunakul P, Suesiritumrong C, Angthong C, Chernchujit B. Validity and Reliability of Thai Version of the Foot and Ankle Ability Measure (FAAM) Subjective Form. J Med Assoc Thai. 2015 Jun;98(6):561-7. PMID 26219160
- [Background] Kline, R.B., 2015. Principles and practice of structural equation modeling: Guilford publications. Principles and practice of structural equation modeling: Guilford publications.